CLINICAL TRIAL: NCT04860986
Title: A Repeatability and Reproducibility Study of the EarliPoint™ Device in Pediatric Subjects 16-30 Months of Age
Brief Title: A Repeatability and Reproducibility Study of the EarliPoint™ Device
Acronym: RnR
Status: Completed | Type: Observational
Sponsor: EarliTec Diagnostics, Inc (Industry)
Responsible Party: Sponsor
Other Study IDs: CLN-1001-001
Record Dates: First submitted 2021-04-14; First posted 2021-04-27 (Actual); Last update posted 2023-11-08 (Actual); Status verified 2023-11

CONDITIONS: Autism Spectrum Disorder (ASD)
Keywords: EarliPoint; Pediatric; Diagnosis
MeSH Terms: conditions — Autism Spectrum Disorder; Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: EarliPoint — EarliPoint is a non-invasive diagnostic device for ASD

SUMMARY:
The study is a prospective randomized repeatability and reproducibility (R&R) study of the EarliPoint DeviceTM in pediatric subjects 16-30 months of age. The study will enroll subjects who are both clinically-positive and clinically-negative for ASD.

The study will be conducted at a single center in the US. The Study consists of a screening period in order to review the subject's medical history to determine subject eligibility, followed by a device administration period during which subjects will undergo testing with the EarliPoint Devices and Expert Clinician Diagnosis (ECD) procedures to determine if they are clinically-positive or clinically-negative for ASD.

DETAILED DESCRIPTION:
Subjects will undergo testing with the same two (2) devices, with one (1) testing session per device per subject, with each testing session yielding three (3) measurements per endpoint per subject, for a total of six (6) measurements per endpoint for each subject enrolled. The order in which the subjects receive testing with each device will be randomized so that the same device is not always used first or last for each subject.

The primary objectives of this study are to quantify the repeatability variability and reproducibility variability of all of the EarliPoint device's continuous valued outputs: the underlying continuous score used to classify patients into the binary diagnostic classification of either clinically-positive or clinically-negative for autism spectrum disorder (ASD) as well as each of the three EarliPoint Device severity scores (the social disability index, verbal ability index, and nonverbal ability index).

The secondary objectives of this study are to quantify the repeatability and reproducibility variability in producing each of the three EarliPoint Device severity scores: the social disability index, verbal ability index, and nonverbal ability index.

ELIGIBILITY:
Inclusion Criteria:

* Children between 16 and 30 months of age.
* No acute illnesses by physical observation.
* Normal or corrected-to-normal vision, and normal or corrected-to-normal hearing.
* Communicate meaningfully with patent in English, and the principal investigator /the study team.
* Parent or legal guardian is able to read and understand the Informed Consent Form.
* Parent voluntarily provides written informed consent.

Exclusion Criteria:

* Genetic disorders (e.g., Fragile X, Williams Syndrome, Tuberous Sclerosis, muscular Dystrophy, Neurofibromatosis, Down Syndrome).
* History or presence of a clinically significant medical disease or a mental state that might confound the study result as assessed by the investigator, such as severe hearing or visual impairment; or uncontrolled epilepsy or seizure disorder, et al.
* Acute exacerbations of chronic illnesses likely to prevent successful data collection.
* Receiving therapies that may affect vision.
* Therapies that may affect the ability to focus.
* Known allergies or sensitivity to the plastic, leather, or metal components.
* Unable or unwilling to sit in a child safety seat.
* Use of any investigational drug, therapies or diagnostic device within the past 14 days.

Ages: 16 Months to 30 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Toddlers and young children will be enrolled in this study, as the aim of this research is to examine repeatability of eye-tracking measures in children aged 16-30 months. Precautions will be taken when working with young children. Our clinicians and research staff are well trained and experienced in working with children and families with some level of anxiety.
  All subject's parent or legal guardian will be consented to the study. No protocol-specific procedures, including screening, will be performed until the parent has signed and dated the consent form. Subjects will also satisfy the inclusion and exclusion criteria in order to be enrolled in the study.
Sampling Method: Non-Probability Sample
Enrollment: 45 (Actual)
Dates: Start 2021-05-07 (Actual); Primary Completion 2021-11-17 (Actual); Study Completion 2021-11-17 (Actual)

PRIMARY OUTCOMES:
The EarliPoint Device repeatability | Anticipated in about 6 months
  EarliPoint Device repeatability agreement in producing binary diagnostic outcomes (clinically-positive or negative for ASD) between multiple measurements per subject conducted with the same device (i.e., intra-device agreement);classification of either clinically-positive or clinically-negative for autism spectrum disorder (ASD) as well as each of the three EarliPoint Device severity scores (the social disability index, verbal ability index, and nonverbal ability index).
The EarliPoint Device reproducibility | Anticipated in about 6 months
  EarliPoint Device reproducibility agreement in producing binary diagnostic outcomes (clinically-positive or negative for ASD) between single measurements per subject conducted with multiple devices (i.e., inter-device agreement);
The repeatability variance of the underlying EarliPoint Device | Anticipated in about 6 months
  Repeatability variance of the underlying EarliPoint Device ASD presence metric (this metric is a continuous score underlying the binary diagnostic outcome: values less than or equal to 0 indicate a patient has ASD [clinically-positive], values greater than 0 indicate a patient does not have ASD [clinically-negative]);
The reproducibility variance of the underlying EarliPoint Device | Anticipated in about 6 months
  reproducibility variance of the underlying EarliPoint Device ASD presence metric (this metric is a continuous score underlying the binary diagnostic outcome: values less than or equal to 0 indicate a patient is ASD positive, values greater than 0 indicate a patient is ASD negative).

CONTACTS AND LOCATIONS:
Overall Officials: Sew-Wah Tay, Study Chair — EarliTec Diagnostics, Inc
Locations (1):
- Emory University, Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: No
There is no plan to share individual participant data (IPD) to other researchers.

REFERENCES:
- [Background] Jones W, Klaiman C, Richardson S, Lambha M, Reid M, Hamner T, Beacham C, Lewis P, Paredes J, Edwards L, Marrus N, Constantino JN, Shultz S, Klin A. Development and Replication of Objective Measurements of Social Visual Engagement to Aid in Early Diagnosis and Assessment of Autism. JAMA Netw Open. 2023 Sep 5;6(9):e2330145. doi: 10.1001/jamanetworkopen.2023.30145. PMID 37669054
- [Background] Jones W, Klaiman C, Richardson S, Aoki C, Smith C, Minjarez M, Bernier R, Pedapati E, Bishop S, Ence W, Wainer A, Moriuchi J, Tay SW, Klin A. Eye-Tracking-Based Measurement of Social Visual Engagement Compared With Expert Clinical Diagnosis of Autism. JAMA. 2023 Sep 5;330(9):854-865. doi: 10.1001/jama.2023.13295. PMID 37668621
- See also: EarliPoint Evaluation for Autism Spectrum Disorder — https://www.earlitecdx.com/solutions/